CLINICAL TRIAL: NCT05250570
Title: Distress Tolerance vs. Relaxation Therapy for Benzodiazepine Discontinuation in Patients Receiving Opioid Agonist Therapy
Brief Title: Distress Tolerance for Benzodiazepine Discontinuation
Acronym: DT-BD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with recruitment
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Tae Woo Park, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21110078; 7K23DA044321-06 (NIH)
Record Dates: First submitted 2022-01-31; First posted 2022-02-22 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distress Tolerance - Benzodiazepine Discontinuation (DT-BD) (Experimental): This psychosocial treatment intervention uses a combination of interoceptive exposure therapy and elements of acceptance and commitment therapy (ACT) and psychoeducation about benzodiazepine use in OAT.
  Interventions: Behavioral: Distress Tolerance - Benzodiazepine Discontinuation (DT-BD)
- Relaxation Therapy (Active Comparator): The relaxation therapy control condition involves psychoeducation about benzodiazepine use in OAT and progressive muscle-relaxation training.
  Interventions: Behavioral: Relaxation Therapy

INTERVENTIONS:
Behavioral: Distress Tolerance - Benzodiazepine Discontinuation (DT-BD) — This psychosocial treatment intervention uses a combination of interoceptive exposure therapy and elements of acceptance and commitment therapy (ACT) to assist individuals in tolerating benzodiazepine withdrawal symptoms and teaching skills to prevent relapse to benzodiazepine use. It will also provide psychoeducation about benzodiazepine use in OAT. Both intervention and control arms will receive identical benzodiazepine discontinuation taper protocols.
  Arms: Distress Tolerance - Benzodiazepine Discontinuation (DT-BD)
Behavioral: Relaxation Therapy — The relaxation therapy control condition involves psychoeducation about benzodiazepine use in OAT and progressive muscle-relaxation training. Both intervention and control arms will receive identical benzodiazepine discontinuation taper protocols.
  Arms: Relaxation Therapy

SUMMARY:
The proposed study is a clinical trial, designed to pilot test a Distress Tolerance-Benzodiazepine Discontinuation (DT-BD) intervention for patients on opioid agonist therapy (OAT) who currently use benzodiazepines versus a Relaxation Therapy (RT) control condition. The DT-BD intervention is an adjunctive psychosocial intervention in people seeking to discontinue (BZD) use.

DETAILED DESCRIPTION:
This study pilot tests a 13-week distress tolerance-based psychosocial intervention paired with a benzodiazepine taper comparing it to a relaxation therapy control condition with the aim of assisting individuals receiving OAT discontinue benzodiazepine use. All participants will receive the same benzodiazepine (BZD) discontinuation protocol. The Distress Tolerance-Benzodiazepine Discontinuation (DT-BD) intervention consists of 13 weeks with 5 weekly therapy sessions prior to a 9-week BZD taper. Some participants may be prescribed non-benzodiazepine medications to treat the underlying conditions for which they were using BZDs [e.g. selective serotonin reuptake inhibitors (SSRI) for anxiety or hypnotics for insomnia]. Data collection will occur at baseline, then weekly for 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Receiving OAT (methadone or buprenorphine) for at least 2 weeks
* Regular BZD use defined by BZD use 3 or more times per week in past month by self-report and positive urine screen at time of recruitment
* Provides permission to contact current BZD prescriber if being prescribed BZDs
* Speaks English
* Wants to discontinue BZD use
* Capacity to provide informed consent

Exclusion Criteria:

* Pregnant, confirmed by urine pregnancy test
* Cognitive impairment, as indicated by Montreal Cognitive Assessment (MoCA): must score at least 26 on the MoCA with a one-point adjustment for individuals with formal education of 12 years or fewer
* Any past month illicit opioid determined by self-report or urine drug test; illicit defined as non-medical use
* Receiving ongoing psychosocial treatment for BZD use disorder
* Uncontrolled seizure disorder (i.e. seizure in prior 90 days), or past BZD withdrawal seizure
* Current suicidality or homicidality
* Current psychotic symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Number of participants who discontinued BZDs at 4-month follow-up | 4-months
  Number of participants with BZD discontinuation defined by no BZD use by self-report during the month prior to 4-month follow-up corroborated by urine testing.
Number of participants who discontinued BZDs at 6-month follow-up | 6-months
  Number of participants with BZD discontinuation defined by no BZD use by self-report during the month prior to 6-month follow-up corroborated by urine testing.

SECONDARY OUTCOMES:
Change in quantity of BZD use | 4- and 6-months
  Change in quantity of BZD used define by past-week BZD use by self-report in diazepam equivalent dose
Change in distress tolerance | 4- and 6-months
  Change in distress tolerance defined by change in Distress Intolerance Index (DII) score from baseline to 6 month follow-up. The DII is a 10-item instrument. Items are rated from 0 (very little) to 4 (very much) and are summed for a total score (range 0-40), with higher scores indicating worse ability to tolerate distress.

OTHER OUTCOMES:
BZD withdrawal symptoms | 4- and 6-months
  BZD withdrawal symptoms will be measured using the Clinical Institute Withdrawal Assessment-Benzodiazepines (CIWA-B). The CIWA-B is a 20-item instrument, to assess severity of benzodiazepine withdrawal, including nausea and vomiting, anxiety, tremor, sweating, auditory disturbances, visual disturbances, tactile disturbances, headache, agitation, and clouding of sensorium. Scores range from 0 to 80, with 1-20 mild withdrawal, 21-40 moderate withdrawal, 41-60 severe withdrawal, and 61-80 very severe withdrawal.
Anxiety symptoms | 4- and 6-months
  Anxiety symptoms will be measured using the Beck Anxiety Inventory (BAI), a 21-item self report inventory for measuring severity of anxiety. The items probe about common symptoms of anxiety that the participant may have experienced in the past week, including numbness, tingling, sweating, and fear. Each item is scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms. The standardized cutoffs are: 0-7: minimal anxiety, 8-15: mild anxiety, 16-25: moderate anxiety, and 26-63: severe anxiety.
Depressive symptoms | 4- and 6-months
  Depressive symptoms will be measured using the Beck Depression Inventory-II, a 21-item self report inventory measuring the severity of depression. The items probe on common symptoms of depression including hopelessness, irritability, guilt, weight-loss, fatigue, or lack of interest in daily activities. Higher total scores indicate more severe depressive symptoms. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Inflexibility or experiential avoidance | 4- and 6-months
  The Acceptance and Action Questionnaire-II will be used to measure inflexibility or experiential avoidance. It is a 7-item self-report measure of psychological inflexibility or experiential avoidance. Each of the 7 items can be rated on a scale of 1 (never true) to 7 (always true) so scores can range from 7 to 49. Higher scores equal greater levels of psychological inflexibility.
Distress tolerance | 4- and 6-months
  Distress tolerance will be assessed with the computerized Mirror Tracing Persistence Task (MTPT-C). It is a computerized version of the original Mirror Tracing Persistence Task in which trace multiple progressively difficult polygons, with participants free to terminate at any point. Distress tolerance is measured by the latency in seconds to task termination. Higher latency indicates greater distress tolerance.
Fear of anxiety symptoms | 4- and 6-months
  Fear of anxiety symptoms will be assessed by the Anxiety Sensitivity Index. It is a 16-item scale with each item rated on a five-point Likert scale ranging from 0 (very little) to 4 (very much). Scores can range from 0 to 64. Higher scores reflect greater fear of anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Tae Woo Park, MD, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - Center for Psychiatric and Chemical Dependency Services (CPCDS), Pittsburgh, Pennsylvania
  - Internal Medicine Recovery Engagement Program (REP), Pittsburgh, Pennsylvania
  - Narcotic Addiction Treatment Program (NATP), Wilkinsburg, Pennsylvania

IPD SHARING:
Plan to Share IPD: No